CLINICAL TRIAL: NCT03508882
Title: Pretarsal Versus Preseptal Botulinum Toxin for Patients With Eyelid Spasm: a Randomized, Triple-blind, Placebo-controlled, Cross-over Clinical Trial
Brief Title: Pretarsal Versus Preseptal Botulinum Toxin for Patients With Eyelid Spasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Marcus M. Marcet, MD, Honorary Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HMRF Project No.: 12133171; Protocol : MMBT; v1.3;1Mar16 (Other: HKU)
Record Dates: First submitted 2018-03-18; First posted 2018-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Blepharospasm; Hemifacial Spasm; Botulinum Toxins, Type A
Keywords: Eyelid; Dystonia; Botulinum injection; Oculoplastics
MeSH Terms: conditions — Blepharospasm; Hemifacial Spasm; Dystonia | interventions — Pharmaceutical Preparations; Botulinum Toxins, Type A; Saline Solution; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preseptal-pretarsal (Active Comparator): The Preseptal-pretarsal group will receive injections of Botulinum Toxin Type A 100Unit/Vial (Product) in the preseptal site (Injection pattern A) and Saline Solution for Injection (placebo control) in the pretarsal site for 2 cycles at 3 months apart. Both groups will crossover and receive the alternative intervention. Hence in the second half of the trial, the Preseptal-pretarsal group will be injected with BtA in Pattern B and Pretarsal-preseptal group will receive Pattern A.
  Interventions: Drug: Botulinum Toxin Type A 100Unit/Vial (Product); Drug: Saline Solution for Injection
- Pretarsal-preseptal (Active Comparator): The Pretarsal-preseptal group will initially receive injections Botulinum Toxin Type A 100Unit/Vial (Product) in the reverse with the intervention at the pretarsal site (Injection pattern B) for 2 cycles at 3 months apart. Groups 1 and 2 will crossover and receive the alternative intervention. Both groups will crossover and receive the alternative intervention. Hence in the second half of the trial, the Preseptal-pretarsal group will be injected with BtA in Pattern B and Pretarsal-preseptal group will receive Pattern A.
  Interventions: Drug: Botulinum Toxin Type A 100Unit/Vial (Product); Drug: Saline Solution for Injection

INTERVENTIONS:
Drug: Botulinum Toxin Type A 100Unit/Vial (Product) — Botulinum Toxin Type A 100Unit/Vial (Product) comes as a dry powder and is routinely reconstituted with Saline Solution for Injection
  Other Names: Botox
Drug: Saline Solution for Injection — The placebo consists of vehicle only. Saline Solution for Injection is the vehicle substance normally used to reconstitute Botulinum Toxin Type A (see 1st Intervention above).
  Other Names: Placebo

SUMMARY:
A triple-masked placebo-controlled trial assessing the efficacy and safety of pretarsal versus preseptal botulinum toxin for patients with eyelid spasm. The investigators hypothesize injection of botulinum toxin into the pretarsal orbicularis oculi muscle will have greater clinical efficacy, better measured quality of life, fewer complications, and better cost effectiveness in comparison to a preseptal pattern of injection.

DETAILED DESCRIPTION:
The study design is a prospective, randomized, triple-blinded placebo controlled crossover trial. A computer-generated list of random numbers will be used for allocation of patients. The patients, treating physicians, and outcome assessors will be masked to the contents of the Botulinum Toxin Type A (BtA) and placebo syringe injections. The placebo will consist of vehicle only, which is the same sterile normal 0.9% saline used in reconstitution of the BtA. At month 6, each group will crossover and receive the alternative intervention. The primary outcome measure (JRS severity) will be the change as measured 1 month after the second cycle of each intervention. Secondary outcome measures include the TWSTRS (clinical response), Blepharospasm Disability Index (BSDI), CDQ-24 (quality of life), VAS (pain), and GAS (global) scores and incidence of side effects. The investigators plan to compare the outcome measures between groups with linear mixed models allowing for the crossover design.

Data will be collected at each of the injection visits and at both of the clinical activity visits. The data will be processed by the research assistant and analysed by the project biostatistician. The investigators plan to compare the primary (JRS) and secondary outcome measures (TWSTRS, BSDI, CDQ-24, VAS, and GAS scores) between the Preseptal-pretarsal (Group 1) and the Pretarsal-preseptal (Group 2) allowing for the crossover design. Specifically, the investigators will use a 2-sample t-test to compare all values of the JRS in group 1 with all the values of the JRS in group 2. This will allow the investigators to determine whether carryover effects are present, and the investigators have specified a 3-month washout period between the first and second round of injections to minimise the chance of carryover effects. If carryover effects are present, the investigators will allow for these in further analysis. The investigators will then use linear mixed models to estimate the difference between the two interventions, allowing for the repeated measures, and if necessary for carryover effects. In secondary analyses, the investigators will evaluate the proportion of patients with relief of spasm, improvement in quality of life, and incidence of side effects, including eyelid ptosis measurements between the two interventions, using logistic regression. P values of 0.05 or less will be considered statistically significant. All analyses will be conducted under the principle of Intention to Treat, using multiple imputation to account for any missing data and to include all randomized patients in analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years-of-age
* Clinical diagnosis eyelid dystonia, consisting of either blepharospasm or hemifacial spasm
* Patient wish to have treatment with botulinum toxin type A (BtA).

Exclusion Criteria:

* Patients unable to express their symptoms or history to the extent that they are not able to complete the study questionnaires, such as those suffering from dementia.
* Existence of potential contraindications to BtA treatment:

  * Pregnancy
  * Breastfeeding
  * Prior allergic reaction
  * Active infection or inflammation in the treatment area
  * Neuromuscular and peripheral neuropathic disease
  * Concomitant aminoglycoside therapy
* Patients with poor or unstable general health with activities of daily living severely affected by non-dystonia confounding factors, such as hospitalized or bed bound patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Jankovic Rating Scale (JRS) | The videos will be taken at the clinical activity visits (C1 and C2) will be scheduled for months 4 and 10. The primary outcome measure will consist of the change from C1 to C2.
  The severity of the patient's spasm employing the widely used JRS scale. The JRS is scored between 0 and 4 (0 = no spasm, 1 = mild, barely noticeable, 2 = mild, without functional impairment, 3 = moderate spasm, moderate functional impairment, 4 = severe incapacitating spasm). The JRS will be scored independently by two graders from a video clip of approximately 30-60 seconds in duration. Differences between the 2 scores will be arbitrated by a third reviewer.

SECONDARY OUTCOMES:
Toronto (TWSTRS) | C1 and C2 will take place at months 4 and 10.
  TWSTRS instrument measuring clinical response. Scored between -1 and 5 (-1 = worse, 0 = no benefit, 1 = minimal or equivocal reduction in spasm, 2 = mild response with some reduction in spasm, 3 = moderate response with some reduction in spasm, 4 = marked reduction of spasm but spasm still present, 5 = major improvement with little or no residual spasm). The change between the 2 clinical activity visits (C1-C2) will be assessed.
Blepharospasm Disability Index (BSDI) | C1 and C2 will take place at months 4 and 10.
  Measure of disability. The change between the 2 clinical activity visits (C1-C2) will be assessed.
Craniocervical Dystonia Questionnaire (CDQ-24) | C1 and C2 will take place at months 4 and 10.
  Measure of quality of life. The change between the 2 clinical activity visits (C1-C2) will be assessed.
Global Assessment Scale (GAS) | C1 and C2 will take place at months 4 and 10.
  To assess the overall status of the patient's disease. The GAS is determined by asking the patient the percentage of function the patient is experiencing. The analogue instrument ranges from "Free of complaints" on the left side to "Suffering extremely" on the right side of a line. Patients self-rate by marking where on the line best represents their current condition. The line measures 100 millimeters long. The mark is measured and the value recorded, ranging from 0 (Free of complaints) to 100 (Suffering extremely). Thus a lower value represents a better outcome.
  The change between the 2 clinical activity visits (C1-C2) will be assessed.
Visual analogue scale (VAS) for pain | Measured at each injection visit (months 0, 3, 6, and 9).
  VAS (range 0-10, no pain = 0, unbearable pain = 0) will be used to assess. The change between the 2 clinical activity visits (C1-C2) will be assessed.
  patients' perception of pain for each of the 2 injections patterns
Ptosis monitoring | C1 and C2 will take place at months 4 and 10.
  Specifically, cropped photographs of both eyelids will be analysed using ImageJ (National Institutes of Health, USA). The Margin-Reflex-Distance 1 (MRD1) measurements will be calculated using the ImageJ software's line tool to capture the height of the upper eyelid and evaluate and quantify the development of any ptosis complications. The change between the 2 clinical activity visits (C1-C2) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus M Marcet, MD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jankovic J. Blepharospasm with basal ganglia lesions. Arch Neurol. 1986 Sep;43(9):866-8. doi: 10.1001/archneur.1986.00520090006004. No abstract available. PMID 3741202
- [Background] Dutton JJ, Fowler AM. Botulinum toxin in ophthalmology. Surv Ophthalmol. 2007 Jan-Feb;52(1):13-31. doi: 10.1016/j.survophthal.2006.10.003. PMID 17212988
- [Background] Czyz CN, Burns JA, Petrie TP, Watkins JR, Cahill KV, Foster JA. Long-term botulinum toxin treatment of benign essential blepharospasm, hemifacial spasm, and Meige syndrome. Am J Ophthalmol. 2013 Jul;156(1):173-177.e2. doi: 10.1016/j.ajo.2013.02.001. Epub 2013 Mar 28. PMID 23541393
- [Background] Harrison AR, Erickson JP, Anderson JS, Lee MS. Pain relief in patients receiving periocular botulinum toxin A. Ophthalmic Plast Reconstr Surg. 2008 Mar-Apr;24(2):113-6. doi: 10.1097/IOP.0b013e31816386e1. PMID 18356715
- [Background] Hilker R, Schischniaschvili M, Ghaemi M, Jacobs A, Rudolf J. Health related quality of life is improved by botulinum neurotoxin type A in long term treated patients with focal dystonia. J Neurol Neurosurg Psychiatry. 2001 Aug;71(2):193-9. doi: 10.1136/jnnp.71.2.193. PMID 11459891
- [Background] Muller J, Wissel J, Kemmler G, Voller B, Bodner T, Schneider A, Wenning GK, Poewe W. Craniocervical dystonia questionnaire (CDQ-24): development and validation of a disease-specific quality of life instrument. J Neurol Neurosurg Psychiatry. 2004 May;75(5):749-53. doi: 10.1136/jnnp.2003.013441. PMID 15090572
- [Background] Hall TA, McGwin G Jr, Searcey K, Xie A, Hupp SL, Owsley C, Kline LB. Health-related quality of life and psychosocial characteristics of patients with benign essential blepharospasm. Arch Ophthalmol. 2006 Jan;124(1):116-9. doi: 10.1001/archopht.124.1.116. PMID 16401794
- [Background] Jankovic J, Schwartz K, Donovan DT. Botulinum toxin treatment of cranial-cervical dystonia, spasmodic dysphonia, other focal dystonias and hemifacial spasm. J Neurol Neurosurg Psychiatry. 1990 Aug;53(8):633-9. doi: 10.1136/jnnp.53.8.633. PMID 2213039
- [Background] Thenganatt MA, Fahn S. Botulinum toxin for the treatment of movement disorders. Curr Neurol Neurosci Rep. 2012 Aug;12(4):399-409. doi: 10.1007/s11910-012-0286-3. PMID 22661378
- [Background] Huang W, Foster JA, Rogachefsky AS. Pharmacology of botulinum toxin. J Am Acad Dermatol. 2000 Aug;43(2 Pt 1):249-59. doi: 10.1067/mjd.2000.105567. PMID 10906647
- [Background] Harrison AR. Chemodenervation for facial dystonias and wrinkles. Curr Opin Ophthalmol. 2003 Oct;14(5):241-5. doi: 10.1097/00055735-200310000-00003. PMID 14502050
- [Background] Costa J, Espirito-Santo C, Borges A, Ferreira JJ, Coelho M, Moore P, Sampaio C. Botulinum toxin type A therapy for blepharospasm. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD004900. doi: 10.1002/14651858.CD004900.pub2. PMID 15674969
- [Background] Aramideh M, Ongerboer de Visser BW, Brans JW, Koelman JH, Speelman JD. Pretarsal application of botulinum toxin for treatment of blepharospasm. J Neurol Neurosurg Psychiatry. 1995 Sep;59(3):309-11. doi: 10.1136/jnnp.59.3.309. PMID 7673963
- [Background] Jankovic J. Pretarsal injection of botulinum toxin for blepharospasm and apraxia of eyelid opening. J Neurol Neurosurg Psychiatry. 1996 Jun;60(6):704. doi: 10.1136/jnnp.60.6.704. No abstract available. PMID 8648354
- [Background] Albanese A, Bentivoglio AR, Colosimo C, Galardi G, Maderna L, Tonali P. Pretarsal injections of botulinum toxin improve blepharospasm in previously unresponsive patients. J Neurol Neurosurg Psychiatry. 1996 Jun;60(6):693-4. doi: 10.1136/jnnp.60.6.693-a. No abstract available. PMID 8648343
- [Background] Cakmur R, Ozturk V, Uzunel F, Donmez B, Idiman F. Comparison of preseptal and pretarsal injections of botulinum toxin in the treatment of blepharospasm and hemifacial spasm. J Neurol. 2002 Jan;249(1):64-8. doi: 10.1007/pl00007849. PMID 11954870
- [Background] Albanese A, Sorbo FD, Comella C, Jinnah HA, Mink JW, Post B, Vidailhet M, Volkmann J, Warner TT, Leentjens AF, Martinez-Martin P, Stebbins GT, Goetz CG, Schrag A. Dystonia rating scales: critique and recommendations. Mov Disord. 2013 Jun 15;28(7):874-83. doi: 10.1002/mds.25579. PMID 23893443
- [Background] Wabbels B, Jost WH, Roggenkamper P. Difficulties with differentiating botulinum toxin treatment effects in essential blepharospasm. J Neural Transm (Vienna). 2011 Jun;118(6):925-43. doi: 10.1007/s00702-010-0546-9. Epub 2011 Jan 9. PMID 21221669
- [Background] Wabbels B, Roggenkamper P. Botulinum toxin in hemifacial spasm: the challenge to assess the effect of treatment. J Neural Transm (Vienna). 2012 Aug;119(8):963-80. doi: 10.1007/s00702-011-0762-y. Epub 2012 Jan 10. PMID 22231846
- [Background] Sarifakioglu N, Sarifakioglu E. Evaluating effects of preservative-containing saline solution on pain perception during botulinum toxin type-a injections at different locations: a prospective, single-blinded, randomized controlled trial. Aesthetic Plast Surg. 2005 Mar-Apr;29(2):113-5. doi: 10.1007/s00266-004-0062-0. Epub 2005 Apr 14. PMID 15815811
- [Background] Jankovic J, Kenney C, Grafe S, Goertelmeyer R, Comes G. Relationship between various clinical outcome assessments in patients with blepharospasm. Mov Disord. 2009 Feb 15;24(3):407-13. doi: 10.1002/mds.22368. PMID 19053054
- [Background] Marcet MM, Lemke BN, Greenwald MJ, Fountain TR, Roth S, Dubovy SR. Eyelid eversion for visualisation of the upper eyelid lamellae: an anatomical cadaver study. Br J Ophthalmol. 2011 Oct;95(10):1376-8. doi: 10.1136/bjophthalmol-2011-300020. Epub 2011 Jul 11. PMID 21746734
- [Background] Marcet MM, Meyer DR, Greenwald MJ, Roth S, Selva D. Proximal tarsal attachments of the levator aponeurosis: implications for blepharoptosis repair. Ophthalmology. 2013 Sep;120(9):1924-9. doi: 10.1016/j.ophtha.2013.02.012. Epub 2013 Apr 16. PMID 23601804
- See also: General information about eyelid spasms and treatment — https://www.asoprs.org/eyelid-spasms